CLINICAL TRIAL: NCT03556267
Title: Role of Beta Trace Protein Assay During Spinal Anesthesia of Cesarean Section
Brief Title: Regional Anesthesia of Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Ali Abdelhaleem Abdelrahman, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ATC 2030
Record Dates: First submitted 2018-05-19; First posted 2018-06-14 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Anesthesia, Obestetric

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spinal needle 27 gauqge (Other): It is a device used to penetrate the dura to take CSF sample before injecting the drugs used for spinal anesthesia for cesarean section.
  Interventions: Device: spinal needle
- spinal needle 25 gauage (Other): It is a device used to penetrate the dura to take CSF sample before injecting the drugs used for spinal anesthesia for cesarean section.
  Interventions: Device: spinal needle

INTERVENTIONS:
Device: spinal needle — It is a spinal needle with 'QUINCKE' Bevel. It is inserted in the lumbar region at the inter-space L4-L5, L4-L3 ,or L3-L2 lumber spaces, while the patient is put in the sitting position then CSF sample is taken then 2.5 ml of a local anesthetic(0.5 ml of 25 ug fentanyl and 2 ml of 8 mg heavy bupivacaine) is given intrathecal then the needle is withdrawn.

SUMMARY:
Beta trace protein assay is an indicator of post-spinal CSF leak that predicts the degree of post-spinal headache.

DETAILED DESCRIPTION:
Beta trace protein is specific for CSF only and it is a quantitative analytic test.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* free medical history.
* free obstetric history.

Exclusion Criteria:

* high risk pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-02-14 (Actual)

PRIMARY OUTCOMES:
CSF sample: serum sample | One year
  After insertion of an intravenous line 4 ml serum will be collected, then 0.5 ml CSF sample will be collected after insertion of the dura by the selected spinal needle before injecting the anesthetic drugs used for spinal anesthesia. Beta trace protein assay will be measured through ELISA technique in both CSF and serum samples and the ratio will be calculated and measured. This ratio will be measured for the three arms aiming at the comparison between the three devices regarding the CSF : Serum ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- Abdelrahman, Cairo, Egypt